CLINICAL TRIAL: NCT04928950
Title: Safety of Oral Activated Charcoal and Its Effect on the Gut Microbiome In Patients With Lung Cancer Undergoing Transcervical Extended Mediastinal Lymphadenectomy (TEMLA)
Brief Title: Charcoal in Lung Cancer Patients Undergoing TEMLA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of logistic challenges and lack of product among other factors, we decided to completely withdrawn this study.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021LS022
Record Dates: First submitted 2021-06-04; First posted 2021-06-16 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Activated charcoal; Gut microbiome; TEMLA
MeSH Terms: conditions — Lung Neoplasms; Anthrax | interventions — Charcoal

STUDY DESIGN:
Intervention Model Description: 15 adults undergoing TEMLA enrolled in a 12-month period.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adults undergoing TEMLA (Experimental): Adults undergoing TEMLA (Transcervical Extended Mediastinal Lymphadenectomy) take Oral Activated Charcoal (OAC) dissolved in apple juice a night before the surgery
  Interventions: Drug: Activated charcoal

INTERVENTIONS:
Drug: Activated charcoal — Activated Charcoal, Powder, USP is carbon that has been treated to create low-volume pores that increase the area available for chemical reactions and adsorption. The most common pharmaceutical uses of activated charcoal is as a purification agent and antitoxin. All Spectrum Chemical USP products are manufactured, packaged and stored under current Good Manufacturing Practices (cGMP) per 21CFR part 211 in FDA registered and inspected facilities.
  Other Names: Medical grade AC, "Activated Charcoal Powder, USP", activated carbon

SUMMARY:
This proof-of-concept study serves as the preliminary step to prove safety of oral activated charcoal (OAC) in patients with solid tumors before moving to a hematologic malignancy patient population.

DETAILED DESCRIPTION:
TEMLA (Transcervical Extended Mediastinal Lymphadenectomy) is a procedure for mediastinal lymph node sampling to stage patients with lung cancer. All patients receive a dose of IV antibiotic pre-procedure to prevent infection. The concept of the proposed study is to protect the gut microbiome against detrimental effects of the antibiotic using oral activated charcoal as a potent adsorbent with no absorption. Oral activated charcoal (OAC) binds to the fraction of IV antibiotic that reaches the lumen of the gut without interfering with its desired systemic effects. The conceptual goal is to prevent dysbiosis by protecting the gut microbiome. Dysbiosis is the leading cause of C. difficile infection and a number of other adverse clinical outcomes such as antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed diagnosis of lung cancer (non-small cell lung cancer, small-cell lung cancer or neuroendocrine tumor) for which a standard of care Transcervical Extended Mediastinal Lymphadenectomy (TEMLA) is planned
* Planned pre-procedural IV antibiotic. The choice of antibiotic type is up to the treatment physician(s)
* Able to safely hold all oral medications on the day of surgery and the day after to ensure the absorption of such drugs is not affected due to charcoal ingestion the night before surgery
* 18 years of age or older
* Able to provide written consent prior to any research related activities

Exclusion Criteria:

* Current pregnancy or breastfeeding (SOC pre-TEMLA testing/assessment)
* Any current diagnosed disease with known involvement of the gastrointestinal tract
* Known allergy to oral activated charcoal
* CTCAE v 5 Dysphagia Grade 2 (symptomatic and altered eating/swallowing) or greater
* Known risk of aspiration based on history or current complaints
* Gastrointestinal procedures within 2 weeks before or (planned) after TEMLA
* Systemic antibiotic use within 8 weeks before planned TEMLA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who are free from analgesics within 3 days of TEMLA | 3 days after surgery
  The duration of analgesic medication use after a standard of care Transcervical Extended Mediastinal Lymphadenectomy (TEMLA) is observed and the number of patients who are free from analgesics is reported

SECONDARY OUTCOMES:
Number of patients experiencing gastrointestinal adverse events | 5 days after surgery
  Incidence of gastrointestinal AEs (nausea, vomiting, abdominal pain, bloating) within 5 days after ingesting charcoal
Number of patients with C. difficile infection | 4 weeks after surgery
  Incidence of C. difficile infection within 4 weeks after TEMLA
Characterization of changes in microbiome diversity | pre-surgery and through study completion, 21-35 days after surgery
  Stool microbiome diversity will be determined by 16S rRNA gene sequencing of samples. Analyses will include alpha and beta diversity, descriptive microbiota composition at the genus level, and comparing these indices between pre- and post- samples.
Characterization of changes in microbiome composition | pre-surgery and through study completion , 21-35 days after surgery
  Stool microbiome composition will be determined by 16S rRNA gene sequencing of samples.

CONTACTS AND LOCATIONS:
Overall Officials: Armin J Rashidi, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota